CLINICAL TRIAL: NCT01162837
Title: An Evaluation of the Safety and Effectiveness of the BEAM Device in the Treatment of Mild-to-moderate Acne
Brief Title: Safety & Effectiveness of the BEAM Device in Mild-to-moderate Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Aesthetic Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OAT-0110
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Other): All subjects are enrolled in this arm and will use the BEAM device on one side of the face and the other side of the face will be the control
  Interventions: Device: BEAM device

INTERVENTIONS:
Device: BEAM device — A red/blue LED device for the treatment of acne

SUMMARY:
This study will determine if the use of the BEAM device reduces the signs and symptoms of mild-to-moderate acne.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 years or older of either gender and of any racial/ethnic group.
2. At least 8 acne inflammatory lesions (see section 9) in the treatment and control areas.
3. Presence of clinically-evident facial acne of mild-to-moderate severity (score 2-4 on the Global Acne Severity Scale, see below)
4. Subjects must be in generally good health.
5. Subjects must be able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. Oral retinoid use within six months of entry into the study.
2. Systemic acne therapies (oral antibiotics) within 2 weeks of entry into the study.
3. Topical acne therapies (retinoids, antibiotics) within 1 week of entry into the study.
4. Microdermabrasion or superficial chemical peels at the site to be treated within 2 months of entry into the study.
5. Subjects with a history of dermabrasion or laser resurfacing at the site to be treated.
6. Use of topical lipid absorbing substances (Clinac AC) within 1 week of entry into the study.
7. Non-compliant subjects.
8. Subjects with a significant medical history or concurrent illness/condition which the investigator(s) feel is not safe for study participation.
9. Subjects using alcohol-based topical solutions or "exfoliating" agents within 1 week of entry into the study.
10. Subjects with a history of very frequent herpes simplex infections of the face or with clinical evidence of active herpes simplex infections.
11. Pregnant or nursing females.
12. Subjects with known photosensitivity disorders felt by the investigators to preclude safe inclusion in the study.
13. Subjects who have a history of significant post-inflammatory hyperpigmentation at the sites of acne lesions.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Reduction in inflammatory lesion count | 8 weeks
  Reduction in the number of inflammatory acne lesions on one side of the face after 8 weeks of treatment.

SECONDARY OUTCOMES:
Global Acne Severity Score | 8-weeks
  Reduction in the Global Acne Severity Score at 8-weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ben Ehst, MD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Baumann Cosmetic & Research Institute, Miami Beach, Florida
  - Grekin Skin Institute, Warren, Michigan
  - Oregon Dermatology & Research Institute, Portland, Oregon